CLINICAL TRIAL: NCT01912157
Title: Couples Coping With Multimorbidity: Does Solitary Expressive Writing Foster Psycho-social Adaptation?
Brief Title: Couples Coping With Multiple Chronic Medical Conditions
Acronym: GUGKS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: KEK-ZH 2013-0009_GUGKS
Record Dates: First submitted 2013-07-24; First posted 2013-07-30 (Estimated); Last update posted 2018-12-31 (Actual); Status verified 2018-12

CONDITIONS: Chronic Disease; Illness Behavior
MeSH Terms: conditions — Chronic Disease; Illness Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No Intervention (Placebo Comparator): The control condition are 3 sessions writing about individual time-management (placebo).
  Interventions: Behavioral: Expressive Writing
- Expressive Writing (Active Comparator): The intervention consists in 3 self-applied solitary written disclosure sessions (expressive writing).
  Interventions: Behavioral: Expressive Writing

INTERVENTIONS:
Behavioral: Expressive Writing — The intervention consists in 3 self-applied solitary written disclosure sessions (expressive writing)

SUMMARY:
Handling of complex health situations (as defined by multimorbidity) in partnership: communication between romantic partners; subjective illness perception; coping with stressful experiences due to multimorbidity.

Intervention : Expressive Writing about subjective illness perception vs. Writing about individual Time-Management Primary Endpoint: subjective Health (e.g. SF 12 questionnaire) Secondary Endpoints: Psychosocial Adjustments (Depression, somatic symptoms, quality of partnership and others)

DETAILED DESCRIPTION:
Coping in complex health situations (as defined by multimorbidity) and the role of relationship processes for psycho-social adaption: The study investigates interpersonal emotion regulation, disclosure, and illness perceptions in couples with a multimorbid patient. The intervention consists in 3 self-applied solitary written disclosure sessions (expressive writing), the control condition are 3 sessions writing about individual time-management (placebo).

Primary endpoint: subjective health (SF 12 questionnaire) Secondary endpoint: psychosocial adjustments (depression, positive and negative affect, somatic symptoms, adjustment disorder, marital satisfaction, sleep quality)

ELIGIBILITY:
Inclusion criteria:

* Age 18 or older
* multimorbid condition (two or more chronic medical conditions)
* patients living with romantic partner
* very good oral and written command in German
* written consent for participation by patient and partner

Exclusion criteria:

* Pregnancy
* Mini Mental State less than 26
* Substance Abuse
* Patients in Palliative Situation
* Patients isolated due to infectious diseases
* Patients participating in other clinical trials within the last 4 weeks before inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2013-07; Primary Completion 2017-04-01 (Actual); Study Completion 2018-12-28 (Actual)

PRIMARY OUTCOMES:
Subjective health (SF-12) | 3 months

SECONDARY OUTCOMES:
Psychosocial adjustments | 3 months
  depression, positive and negative affect, somatic symptoms, adjustment disorder, marital satisfaction, sleep quality

CONTACTS AND LOCATIONS:
Overall Officials: Lukas Zimmerli, MD, Principal Investigator — University Hospital Zurich, Internal Medicine
Locations (1):
- University Hospital Zurich, Internal Medicine, Zurich, Canton of Zurich, Switzerland